CLINICAL TRIAL: NCT05674526
Title: A Phase 1b Study of WU-NK-101 in Combination With Cetuximab for Advanced and/or Metastatic Colorectal Cancer (CRC) and Advanced and/or Metastatic Squamous Cell Carcinoma of the Head and Neck (SCCHN)
Brief Title: A Phase 1b Study of WU-NK-101 in Combination With Cetuximab
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Wugen, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WUN101-02
Record Dates: First submitted 2022-12-30; First posted 2023-01-06 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Colorectal Cancer Metastatic; Squamous Cell Carcinoma of Head and Neck
Keywords: NK cells; allogeneic NK cells; cetuximab
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Intervention Model Description: In dose expansion patients will be enrolled in 2 parallel, disease specific cohorts to further characterize the safety, tolerability and preliminary anti- tumor activity of WU-NK-101 in combination with cetuximab
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- WU-NK-101 Monotherapy/Cetuximab combo Run-in (Experimental): WU-NK-101 is a non-engineered Natural Killer (NK) cell derived from peripheral blood mononuclear cells (PBMC) that is cytokine-reprogrammed, expanded, and cryopreserved to create an allogeneic enhanced memory-like anti-tumor NK cell therapy product.
  Each 8 week cycle in dose escalation is divided into two 28- days segments. Patients will receive WU-NK-101 (Days 1 and 15) in the first segment and a combination of cetuximab (500mg/m2 on Days 29 and 43) plus WU-NK-101 (Days 30 and 44) in the second segment.
  Interventions: Biological: WU-NK-101 - Dose Escalation; Drug: Cetuximab - Dose Escalation
- WU-NK-101 /Cetuximab Combo (Experimental): Patients will receive cetuximab dosed at 500 mg/m2 on Days 1 and 15, and WU-NK-101 on Days 2 and 16, in each 4-week cycle. Depending on response patients may receive up to 6 cycles of treatment.
  Interventions: Biological: WU-NK-101 - Cohort Expansion; Biological: Cetuximab - Cohort Expansion

INTERVENTIONS:
Biological: WU-NK-101 - Dose Escalation — WU-NK-101 administered on Days 1, 15, 30 and 44
  Arms: WU-NK-101 Monotherapy/Cetuximab combo Run-in
Drug: Cetuximab - Dose Escalation — Cetuximab 500mg/m2 administered on Days 29 and 43
  Arms: WU-NK-101 Monotherapy/Cetuximab combo Run-in
Biological: WU-NK-101 - Cohort Expansion — WU-NK-101 administered on Days 2 and 16
  Arms: WU-NK-101 /Cetuximab Combo
Biological: Cetuximab - Cohort Expansion — Cetuximab 500mg/m2 administered on Days 1 and 15
  Arms: WU-NK-101 /Cetuximab Combo

SUMMARY:
This study is a Phase 1b open-label study designed to characterize the safety, tolerability, and preliminary anti-tumor activity of WU-NK-101 in combination with cetuximab in patients with advanced and/or metastatic CRC (Cohort 1), and in patients with advanced and/or metastatic SCCHN (Cohort 2). The overall study will be comprised of two phases, a Dose Escalation Phase, and a Cohort Expansion Phase.

DETAILED DESCRIPTION:
In the Dose Escalation Phase, up to 12 patients with either advanced and/or metastatic CRC or advanced and/or metastatic SCCHN will be treated with WU-NK-101, alone and in combination with cetuximab, in successive cohorts of 3 to 6 patients using a standard 3 + 3 design. Intra-patient dose escalation is not permitted. Patients may receive up to one 8-week cycle of treatment. Each 8-week cycle is divided into two 28-day segments, (Segments A and B).

During Segment A, only WU-NK-101 (monotherapy) will be administered. Segment A will consist of two doses of WU-NK-101 infused on Day 1 and Day 15. Patients that do not experience a dose limiting toxicity (DLT) will proceed to Segment B.

During Segment B, WU-NK-101 will be administered in combination with cetuximab (combination therapy). WU-NK-101 cells will be administered on Days 30 and 44. Cetuximab will be administered on Days 29 and 43 at 500 mg/m2 (FDA-approved dose).

Once the MTD/MAD is defined in the Dose Escalation Phase, up to 9 additional patients will be enrolled in 2 parallel, disease specific, expansion cohorts (Cohort 1 [patients with CRC] and Cohort 2 [patients with SCCHN]) to further characterize the safety, tolerability, and preliminary anti-tumor activity of WU-NK-101 cells in combination with cetuximab. Patients will receive cetuximab dosed at 500 mg/m2 on Days 1 and 15, and WU-NK-101 on Days 2 and 16, in each 4-week cycle.

At the end of Cycle 2, patients who achieve a partial response (PR) or stable disease (SD) may receive up to 4 additional cycles of treatment of WU-NK-101 cells in combination with cetuximab with disease assessments on Day 28 (+/- 3 days) of each even numbered cycle, for a maximum of 6 cycles.

ELIGIBILITY:
Inclusion Criteria:

Patients must have a histologically confirmed diagnosis of advanced and/or metastatic CRC that has failed or progressed beyond first line or higher line standard of care therapy including bevacizumab combination, cetuximab combination, 5-FU based regimens, or checkpoint inhibitors alone or in combination. Patients must have received all targeted therapies for which they are eligible. Patients may be included in this study regardless of mutation status (e.g., RAS-mutant, wild-type, or unknown status, BRAF V600E, etc.) and EGFR expression.

Or,

Patients must have a histologically confirmed diagnosis of SCCHN that has failed or progressed beyond first or higher line standard of care therapy including cetuximab alone or in combination, checkpoint inhibitors alone and in combination, or regimens containing radiotherapy. Patients may be included in this study regardless of EGFR expression.

Exclusion Criteria:

Experienced toxicities related to prior cetuximab treatment which required permanent discontinuation of cetuximab per the current label.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05-21 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events of WU-NK-101 in combination with cetuximab as assessed by by CTCAE v5 | 24 months
  Safety is based on evaluation of adverse events (AEs) and serious adverse events (SAEs) from the time of consent until the end of the study visit or at the end of treatment visit.
Maximum Tolerated Dose | up to 56 days from first dose
  Maximum tolerated or administered dose of WU-NK-101 in combination with cetuximab

SECONDARY OUTCOMES:
Duration of Response | 24 months
  Time of response to the time of disease relapse, progression or death due to any cause
Overall Response Rate | 24 months
  ORR is defined as the proportion of patients that achieve complete remission (CR) + partial response (PR) using modified Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST 1.1)

CONTACTS AND LOCATIONS:
Overall Officials: Cherry Thomas, MD, Study Director — Wugen, Inc.
Locations (2):
- United States (2):
  - UCSF, San Francisco, California
  - Montefiore Medical Center, The Bronx, New York